CLINICAL TRIAL: NCT03049033
Title: Neurologic Music Therapy for Enhancing Fine Motor Control in Parkinson's Disease
Brief Title: NMT for Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-2308; K01AT009894 (NIH)
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neurologic Music Therapy (NMT) (Experimental): Neurologic Music Therapy is a 5-week intervention using different musical instruments and auditory cues to specifically improve fine motor movements.
  Interventions: Other: Neurologic Music Therapy
- Occupational Therapy (OT) (Active Comparator): Standard of care occupational therapy uses traditional motor training.
  Interventions: Other: Occupational Therapy
- Waitlist Control (No Intervention): Participants assigned to the waitlist-control condition will not immediately receive services. The no-treatment duration for these participants is yoked to the amount of time their respective NMT- and OT-condition participants receive services (5 weeks). After the wait period, these participants will then be randomized to receive either NMT, MST or OT sessions.
- Music Supported Therapy (MST) (Active Comparator): Music Supported Therapy uses musical instruments to train fine motor movements.
  Interventions: Other: Music Supported Therapy

INTERVENTIONS:
Other: Neurologic Music Therapy — Neurologic Music Therapy uses rhythms to change brain activity and function.
  Arms: Neurologic Music Therapy (NMT)
Other: Occupational Therapy — Occupational Therapy uses traditional motor training.
  Arms: Occupational Therapy (OT)
Other: Music Supported Therapy — Music Supported Therapy uses musical instruments to train fine motor movements.
  Arms: Music Supported Therapy (MST)

SUMMARY:
Parkinson's Disease (PD) is defined by characteristic motor symptoms including slow movements, small movements, difficulty with movement initiation and disruptions in timing. Besides gross motor symptoms, fine motor impairments in PD cause difficulties with everyday tasks such as writing, self-care, and fine object manipulation. These activity limitations can lead to disability, social isolation, and a reduced quality of life. In a series of breakthrough studies Michael Thaut and colleagues developed Neurologic Music Therapy (NMT) and found it can address many gross motor impairments and improve gait and balance. Other music therapies such as Music-supported Therapy (MST) have proven motor benefits in stroke patients through movement exercises with musical instruments. However, the pathological basal ganglia (BG) in PD brains leads to a reduced supply of those internally generated movements. In contrast, externally cued movements (eg. via a beat or a rhythm) during NMT sessions are instantaneously entrained to the period of a rhythmic stimulus possibly without involvement of the BG. The underlying idea is that rhythm is the essential component relating music specifically to motor behavior. The mechanism of action is called "rhythmic entrainment" where one system's motion or signal frequency entrains the frequency of another system. The effect of NMT on fine motor function has not been investigated yet. Music activities are important in the lives of many older adults. Notably, the use of music has been associated with increased well-being for older adults, as it fosters social connection and mood regulation. Furthermore, many musical activities have limited physical demands, making them attainable for individuals who are living with mobility impairments or other physical restrictions. Based on the literature and the investigators preliminary studies, the investigators propose to test the efficacy of Neurologic Music Therapy in comparison to Music Supported Therapy and Occupational Therapy (OT) as standard of care on adults in the Parkinson's spectrum. The investigators have defined a working plan using different musical instruments and growing tempo to specifically improve fine motor movements.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 to 85
* Diagnosis of Parkinson's Disease using the UK Brain Bank Criteria
* Fine motor impairments (if available, scores 2 and higher on the UPDRS motor examination part III.23 and 24)
* Medication stable for at least 30 days.

Exclusion Criteria:

* Features suggestive of other causes of parkinsonism, including cerebrovascular disease or history of major head trauma
* Inability to move fingers or hands
* Hoehn and Yahr stage 4 and higher
* Ferrous metal implants which may interfere with the MEG data acquisition and/or be an MRI safety concern
* Dementia
* Participants engaged in other research studies involving music therapies
* Participants whose insurance does not cover Occupational Therapy costs or who have no insurance.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Outcome: Motor 1 (change in the Grooved Pegboard Test) | Baseline and 5 weeks
  First motor outcome will be a change in the Grooved Pegboard Test.
Quality of Life (QOL) Outcome: QOL 1 (change in the 39-Item Parkinson's Disease) | Baseline and 5 weeks
  First QOL outcome will be a change in the 39-Item Parkinson's Disease Questionnaire.
Mechanistic Outcome: Neurophysiology 1 (change in motor beta and gamma power using Magnetoencephalography) | Baseline and 5 weeks
  Our first mechanistic outcome will be a change in cortical motor beta and gamma power using Magnetoencephalography.
Mechanistic Outcome: Neurophysiology 2 (change in auditory-motor functional connectivity using Magnetoencephalography) | Baseline and 5 weeks
  Our second neurophysiology outcome will be a change in auditory-motor functional connectivity using Magnetoencephalography

SECONDARY OUTCOMES:
Clinical Outcome: Motor 2 (change in the Unified Parkinson Disease Rating Scale Part III) | Baseline and 5 weeks
  Secondary motor outcome will be a change in the Unified Parkinson Disease Rating Scale Part III.
Clinical Outcome: Motor 3 (change in the Finger-Thumb opposition from the Neurological Evaluation Scale) | Baseline and 5 weeks
  Secondary motor outcome will be a change in the Finger-Thumb opposition from the Neurological Evaluation Scale.
Quality of Life (QOL) Outcome: QOL 2 (change in the Clinical Global Impression - Improvement Scale) | Baseline and 5 weeks
  Second QOL outcomes will be a change in the Clinical Global Impression - Improvement Scale .
Quality of Life (QOL) Outcome: QOL 3 (change in the Hospital Anxiety and Depression Scale) | Baseline and 5 weeks
  Second QOL outcomes will be a change in the Hospital Anxiety and Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Buard, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available to the scientific community upon request.
  Data sharing will include motor tests, questionnaires and MEG raw data.

REFERENCES:
- [Derived] Buard I, Lattanzio L, Stewart R, Thompson S, Sjoberg K, Hookstadt K, Morrow M, Holden SK, Sillau S, Thaut M, Kluger B. Randomized controlled trial of neurologic music therapy in Parkinson's disease: research rehabilitation protocols for mechanistic and clinical investigations. Trials. 2021 Aug 28;22(1):577. doi: 10.1186/s13063-021-05560-7. PMID 34454592